CLINICAL TRIAL: NCT01204931
Title: Can We Predict Who Has GERD? Systematic Evaluation of Role of pH Monitoring and the Specific Physiologic pH Parameters in Defining GERD, Bravo, Impedence and SISAP
Brief Title: Can We Predict Who Has Gastroesophageal Reflux Disease (GERD)?
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Michael Vaezi, Medical Director, Vanderbilt University
Other Study IDs: GERD SISAP
Record Dates: First submitted 2010-09-13; First posted 2010-09-17 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-09

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: reflux; gastroesophageal reflux disease; GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gastroesophageal Reflux Disease (GERD) Cases: Erosive disease - presence of esophageal mucosal injuries documented endoscopically.
  Non-erosive disease - normal esophagogastroduodenoscopy with symptoms
- Control Group: normal subjects without symptoms of gastroesophageal reflux disease (GERD)

SUMMARY:
Gastroesophageal reflux disease (GERD) is currently defined as "a condition which develops when the reflux of stomach contents causes troublesome symptoms and/or complications". Doctors often diagnose and treat GERD based on symptoms of heartburn and regurgitation. In recent years, the prevalence of partial or non-response to Proton Pump Inhibitors (PPI) has increased resulting in diagnostic testing with esophagogastroduodenoscopy (EGD) or ambulatory pH monitoring. Most patients do not have endoscopic evidence for reflux. Thus, in this group pH monitoring has emerged as an important physiologic test to determine the degree of esophageal acid exposure and to assess the association between patients' persistent symptoms and acid reflux events. The aims of this study are to assess the sensitivity and specificity of symptom associated indices and determine the best parameter for predicting GERD from a list of conventional pH measurement findings.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ages 18 or older
* Presenting to the Vanderbilt GI outpatient clinic with symptoms of GERD
* Undergoing upper endoscopy and wireless pH monitoring (standard of care)
* Erosive disease: presence of esophageal mucosal injuries documented
* Non-erosive disease: normal esophagogastroduodenoscopy (EGD) with symptoms
* Control group: normal subjects without symptoms of GERD

Exclusion Criteria:

* Anti-reflux therapy within 7 days prior to the pH study
* Previous neck, esophagus, or stomach surgery
* Major motility disorders
* Previous neck, esophagus, or stomach cancer or radiations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult subjects presenting to Vanderbilt University Medical Center Gastroenterology outpatient clinic with symptoms consistent with gastroesophageal reflux disease (GERD)
Sampling Method: Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2010-11; Primary Completion 2013-07 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Symptom Index (SI) and Symptom Associated Probability (SAP) | Following esophagogastroduodenoscopy (EGD) and 48-hr-wireless pH monitoring
  Assess the sensitivity and specificity of symptom association indices (SI and SAP)regarding gastroesophageal reflux disease (GERD)
Predicting gastroesophageal reflux disease (GERD) | Following esophagogastroduodenoscopy (EGD) and 48-hr-wireless pH monitoring
  Determine the best parameter for predicting gastroesophageal reflux disease (GERD) from a list of conventional pH measurement findings.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Vaezi, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center GI Outpatient Clinic, Nashville, Tennessee, United States